CLINICAL TRIAL: NCT01651000
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy and Safety of CTAP101 Capsules to Treat Secondary Hyperparathyroidism in Subjects With Stage 3 or 4 Chronic Kidney Disease and Vitamin D Insufficiency
Brief Title: Safety and Efficacy of CTAP101 to Treat Secondary Hyperparathyroidism in Stage 3 or 4 CKD and Vitamin D Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OPKO IP Holdings II, Inc. (Industry)
Responsible Party: Sponsor
Organization: OPKO Health, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTAP101-CL-3001
Record Dates: First submitted 2012-07-23; First posted 2012-07-26 (Estimated); Results first posted 2016-08-17 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2019-12

CONDITIONS: Chronic Kidney Disease; Hyperparathyroidism, Secondary; Vitamin D Deficiency
Keywords: Parathyroid Diseases; Renal Insufficiency; Kidney Failure, Chronic; Hyperparathyroidism, Secondary; Vitamin D; Hyperparathyroidism; Kidney Diseases; Kidney Failure; Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary; Vitamin D Deficiency; Parathyroid Diseases; Renal Insufficiency; Kidney Failure, Chronic; Hyperparathyroidism; Kidney Diseases | interventions — Calcifediol; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CTAP101 30 μg capsules (Active Comparator): 1 CTAP101 30 μg capsule daily at bedtime for 12 weeks, with a possible increase to 2 CTAP101 30 μg capsules daily at bedtime for study duration, if needed (26 weeks total). Subjects not requiring a dose increase after 12 weeks would receive 1 CTAP101 30 μg capsule and one sugar pill (to CTAP101 30 μg capsule) for weeks 13-26.
  Interventions: Drug: CTAP101 30 μg capsules; Other: Sugar pill to CTAP101 30 μg capsules
- Sugar pill to CTAP101 30 μg capsule (Placebo Comparator): 1 sugar pill to CTAP101 30 μg capsule daily at bedtime for 12 weeks, with an increase to 2 sugar pills to CTAP101 30 μg capsules daily at bedtime for weeks 13-26.
  Interventions: Other: Sugar pill to CTAP101 30 μg capsules

INTERVENTIONS:
Drug: CTAP101 30 μg capsules — CTAP101 30 μg capsule taken daily at bedtime.
  Other Names: Calcifediol
  Arms: CTAP101 30 μg capsules
Other: Sugar pill to CTAP101 30 μg capsules — Sugar pill capsule (placebo to CTAP101 30 μg capsule) taken daily at bedtime.
  Other Names: Placebo

SUMMARY:
This study will evaluate the efficacy of CTAP101 Capsules versus placebo in reducing intact parathyroid hormone (iPTH) by at least 30% from pretreatment baseline; safety and tolerability of CTAP101 will also be evaluated

DETAILED DESCRIPTION:
This is a phase 3, multi-center, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of CTAP101 Capsules administered for 26 weeks to treat SHPT in subjects ≥18 years of age with stage 3 or 4 CKD and vitamin D insufficiency. The study will be conducted at approximately 40 sites within the United States (US). Approximately 550 subjects will be screened to randomize approximately 210 eligible subjects, stratified by CKD stage (approximately 105 subjects in each stage) in a 2:1 ratio to receive either CTAP101 Capsules or matching placebo. An Interactive Voice Response System (IVRS) will provide study treatment group assignments using the computer-generated randomization code provided by the IVRS vendor. Subjects will receive an initial daily dose of 1 capsule (CTAP101 Capsules, 30 µg, or matching placebo) for the first 12 weeks. After l2 weeks (visit 8) and per pre-defined criteria, the dose may be increased in a blinded fashion by the IVRS with oversight by an independent medical monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Urinary albumin excretion ≤ 3000 mcg/mg of creatinine
2. Stage 3 or 4 CKD
3. Plasma iPTH: ≥ 85 pg/mL and < 500 pg/mL
4. Serum Ca: ≥ 8.4 mg/dL and < 9.8 mg/dL
5. Serum P: ≥ 2.0 mg/dL and < 5.0 mg/dL
6. Serum 25-hydroxyvitamin D: ≥ 10 ng/mL and < 30 ng/mL.
7. Stable dose of Vitamin D therapy ≤ 1600 IU/day and receiving same dose for at least 2 months

Exclusion Criteria:

1. History of kidney transplant or parathyroidectomy
2. Spot urine calcium:creatinine ratio > 0.2 (>200 mg/g Cr)
3. Current serious illness, such as malignancy, HIV, liver disease, cardiovascular event or hepatitis
4. Currently on dialysis
5. Use of pharmacological dose of ergocalciferol or cholecalciferol (≥ 50,000 IU mcg per month) during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Melnick, MD, Study Director — Opko Renal
Locations (1):
- OPKO Renal, Bannockburn, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted at 44 investigational sites within the US. Subjects were enrolled and treated from 07 September 2012 through 20 July 2014.
Pre-assignment Details: Subjects were stratified by CKD stage and were randomized in a 2:1 ratio to receive a daily 30 μg oral dose of CTAP101 capsules (or matching placebo) for 12 weeks at bedtime. Subjects presenting on a regimen of bone metabolism therapy were to discontinue their prior treatment for at least 28 days' washout (except for bisphosphonates).
Groups:
- CTAP101 30 μg Capsules: 1 CTAP101 30 μg capsule daily at bedtime for 12 weeks, with a possible increase in a blinded fashion to 2 CTAP101 30 μg capsules daily at bedtime for study duration, if needed (26 weeks total). Subjects not requiring a dose increase after 12 weeks would receive 1 CTAP101 30 μg capsule and one sugar pill (to CTAP101 30 μg capsule) for weeks 13-26.
  CTAP101 30 μg capsules: CTAP101 30 μg capsule taken daily at bedtime.
  Sugar pill to CTAP101 30 μg capsules: Sugar pill capsule (placebo to CTAP101 30 μg capsule) taken daily at bedtime.
Period: Overall Study
Arm/Group | Sugar Pill to CTAP101 30 μg Capsule | CTAP101 30 μg Capsules
Started | 72 | 141
Entered Extension Study | 50 | 93
Completed | 62 | 113
Not Completed | 10 | 28
Not completed — Adverse Event | 2 | 8
Not completed — Lost to Follow-up | 3 | 2
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal by Subject | 2 | 10
Not completed — Subject noncompliance | 0 | 3
Not completed — Lack of Efficacy | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Administrative reason | 1 | 0
Not completed — Serum Ca >/= 11.0 mg/dL, repeat confirm | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill to CTAP101 30 μg Capsule | CTAP101 30 μg Capsules | Total
Number analyzed (Participants) | 72 | 141 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (12.74) | 65.1 (10.33) | 64.9 (11.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 71 | 104
  Male | 39 | 70 | 109
Region of Enrollment [Number; unit: participants]
  United States | 72 | 141 | 213

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in the Intent to Treat Population With Decrease in Plasma Intact Parathyroid Hormone (iPTH) of ≥30% From Pre-treatment Baseline Values
Description: Number of subjects in the intent to treat population attaining a mean decrease in plasma intact parathyroid hormone (iPTH) of ≥30% from pre-treatment baseline in the efficacy assessment phase (EAP), referred to as responders.
Time Frame: Approximately 6 months
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Sugar Pill to CTAP101 30 μg Capsule | CTAP101 30 μg Capsules
Number analyzed (Participants) | 72 | 141
participants | 6 | 46
Statistical Analysis 1: Comparison: Sugar Pill to CTAP101 30 μg Capsule vs CTAP101 30 μg Capsules; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Number of Participants in the Per Protocol Population With Decrease in Plasma Intact Parathyroid Hormone (iPTH) of ≥30% From Pre-treatment Baseline Values
Description: Number of subjects in the per protocol population attaining a mean decrease in plasma intact parathyroid hormone (iPTH) of ≥30% from pre-treatment baseline in the efficacy assessment phase (EAP), referred to as responders.
Time Frame: Approximately 6 months
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Sugar Pill to CTAP101 30 μg Capsule | CTAP101 30 μg Capsules
Number analyzed (Participants) | 62 | 115
participants | 5 | 46
Statistical Analysis 1: Comparison: Sugar Pill to CTAP101 30 μg Capsule vs CTAP101 30 μg Capsules; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Subjects in the Intent to Treat Population With Normal Serum Total 25-hydroxyvitamin D
Description: Subjects in the Intent to Treat Population with normal serum total 25-hydroxyvitamin D (>/= 30 ng/dL)
Time Frame: Approximately 6 months
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | Sugar Pill to CTAP101 30 μg Capsule | CTAP101 30 μg Capsules
Number analyzed (Participants) | 72 | 141
participants | 2 | 113
Statistical Analysis 1: Comparison: Sugar Pill to CTAP101 30 μg Capsule vs CTAP101 30 μg Capsules; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Subjects in the Per Protocol Population With Normal Serum Total 25-hydroxyvitamin D
Description: Subjects in the Per Protocol Population with normal serum total 25-hydroxyvitamin D (>/= 30 ng/mL)
Time Frame: Approximately 6 months
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Sugar Pill to CTAP101 30 μg Capsule | CTAP101 30 μg Capsules
Number analyzed (Participants) | 62 | 115
participants | 2 | 110

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Sugar Pill to CTAP101 30 μg Capsule | CTAP101 30 μg Capsules
Serious Adverse Events (participants affected / at risk) | 12/72 | 30/141
Other Adverse Events (participants affected / at risk) | 37/72 | 44/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill to CTAP101 30 μg Capsule (N=72) | CTAP101 30 μg Capsules (N=141)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Arrhyhmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 6 (6)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 5 (5)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal ganglia stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aortic intramural haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill to CTAP101 30 μg Capsule (N=72) | CTAP101 30 μg Capsules (N=141)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 6 (6)
Nausea (Gastrointestinal disorders) | 6 (6) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2)
Oedema peripheral (General disorders) | 5 (5) | 3 (3)
Chest pain (General disorders) | 4 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 10 (10) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Hypertension (Vascular disorders) | 5 (5) | 9 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less